CLINICAL TRIAL: NCT01579435
Title: Thérapeutique expérimentale du Tremblement Essentiel Par la Stimulation Trans-crânienne Par Courant Direct (tDCS) du Cortex cérébelleux et du Cortex Moteur. Etude Exploratoire.
Brief Title: Experimental Therapeutics in Essential Tremor Using Transcranial Direct Current Stimulation
Acronym: ELECTRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C11-37; 2011-A01453-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-04-05; First posted 2012-04-18 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Essential Tremor
Keywords: essential tremor; primary motor cortex; cerebellum; transcranial direct current stimulation; electrophysiology
MeSH Terms: conditions — Essential Tremor | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic tDCS (Experimental): 6 patients with essential tremor
  Interventions: Device: transcranial direct current stimulation
- Physiopathological tDCS (Experimental): 6 patients with essential tremor
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Active stimulation: duration: 20 mn, intensity: 2 mA; localisation : motor cortex or cerebellum; Placebo stimulation: duration: 9 seconds, intensity: 2 mA; localisation : motor cortex or cerebellum;

SUMMARY:
The purpose of this study is to determine whether transcranial direct current stimulation (tDCS) delivered over the motor cortex or the cerebellum can improve essential tremor and to identify the cerebral mechanisms involved in these potential effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 50 years
* Important essential tremor (bilateral postural and/or action tremor since more than one year)
* Normal physical and neurological examination, except for essential tremor
* Insufficient efficiency of usual essential tremor's treatment
* No treatment altering the cortical excitability
* Agreement to use a medically acceptable method of contraception throughout the study for female of childbearing potential

Exclusion Criteria:

* Cervical tremor
* Current neurological or psychiatric illness other than essential tremor
* Individual who is on medication which is known to lower seizure threshold
* Previous history of seizure(s), malaise or current active epilepsy
* Contraindication for MRI or TMS study
* Pregnancy, breast feeding women and women who are of childbearing age and not practicing adequate birth control
* Individual who have MMS ≤ 24/30 or patients legally protected or inability to provide an informed consent
* Simultaneous participation in another clinical trial
* Patients who are not enrolled at social security

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in tremor amplitude on accelerometric recording 10 minutes after the end of tDCS | 10 minutes after the end of tDCS

SECONDARY OUTCOMES:
Change from baseline in tremor amplitude on electromyographic recordings | During tDCS (expected average of 15 minutes), 10 and 60 mn after the end of tDCS
Change from baseline in tremor amplitude on digitized tablet | During tDCS (expected average of 15 minutes), 10 and 60 mn after the end of tDCS
Change from baseline in tremor amplitude on accelerometric recording | During tDCS (expected average of 15 minutes) and 60 minutes after the end of tDCS

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Flamand-Roze, MD, Principal Investigator — Institut du Cerveau et de la Moelle et Fédération de Neurologie de l'Hôpital Pitié-Salpétrière, Paris
Locations (1):
- Institut du Cerveau et de la Moelle, Hôpital Pitié-Salpétrière, Paris, France